CLINICAL TRIAL: NCT02462148
Title: Perineural Steroids for Saphenous Peripheral Nerve Blocks: An Equivalency Dosing Study.
Brief Title: Perineural Steroids for Peripheral Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00032807
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Anesthesia; Anesthesia, Conduction; Anesthesia, Local; Bupivacaine; Dexamethasone; Saphenous; Adductor Canal; Nerve Block; Analgesia; Preanesthetic Medication; Perioperative Period; Peripheral Nerve Block
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Dexamethasone; dexamethasone 21-phosphate; Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 mg Perineural Dexamethasone Group (Experimental): 4 mg of dexamethasone will be included in the saphenous nerve block mixture including 20 ml of 0.25% bupivacaine with 1:400,000 epinephrine. No systemic dexamethasone will be given.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Drug: Epinephrine; Procedure: Saphenous Peripheral Nerve Block
- 1 mg Perineural Dexamethasone Group (Experimental): 1 mg of dexamethasone will be included in the saphenous nerve block mixture including 20 ml of 0.25% bupivacaine with 1:400,000 epinephrine. No systemic dexamethasone will be given.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Drug: Epinephrine; Procedure: Saphenous Peripheral Nerve Block
- Placebo Group (Placebo Comparator): This group will receive only the saphenous nerve block mixture including 20 ml of 0.25% bupivacaine with 1:400,000 epinephrine. Dexamethasone will not be administered to this group systemically or perineural.
  Interventions: Drug: Bupivacaine; Drug: Epinephrine; Procedure: Saphenous Peripheral Nerve Block

INTERVENTIONS:
Drug: Dexamethasone — Used in nerve block mixture
  Other Names: Dexamethasone Sodium Phosphate Injection
  Arms: 1 mg Perineural Dexamethasone Group; 4 mg Perineural Dexamethasone Group
Drug: Bupivacaine — Used in nerve block mixture
  Other Names: Bupivacaine Hydrochloride
Drug: Epinephrine — Used in nerve block mixture
  Other Names: Adrenaline
Procedure: Saphenous Peripheral Nerve Block — Peripheral nerve block.
  Other Names: Adductor Canal Peripheral Nerve Block

SUMMARY:
This study will look at the efficacy of dexamethasone for prolongation of peripheral nerve blocks.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blinded, placebo-controlled trial is to examine if dexamethasone given perineurally as an adjuvant to the nerve block will prolong the time to recovery from sensory nerve block from a saphenous (or adductor canal) nerve block. The primary outcome will be time to resolution of the nerve block as assessed by pinprick over the saphenous nerve distribution. If this primary end point is met, this study will also serve as an equivalency dosing study comparing 1 mg of perineural dexamethasone to 4 mg of perineural dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* elective robotic medial MAKO partial knee arthroplasty
* agreed to a regional anesthesia technique

Exclusion Criteria:

* contraindications to regional anesthesia
* presence of a progressive neurological deficit
* a pre-existing coagulopathy, infection
* insulin and non-insulin dependent diabetes mellitus
* systemic use of corticosteroids within 30 days of surgery
* chronic use of an opioid analgesic (>3 months or a combined total of more than 40 mg Oxycodone equivalents a day)
* pregnancy
* a prior history of an adverse event (for example: psychosis) or an allergy to dexamethasone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl S Henshaw, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Turner JD, Henshaw DS, Weller RS, Jaffe JD, Edwards CJ, Reynolds JW, Russell GB, Dobson SW. Perineural dexamethasone successfully prolongs adductor canal block when assessed by objective pinprick sensory testing: A prospective, randomized, dose-dependent, placebo-controlled equivalency trial. J Clin Anesth. 2018 Aug;48:51-57. doi: 10.1016/j.jclinane.2018.05.009. Epub 2018 May 9. PMID 29753264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
Started | 37 | 36 | 12
Completed | 36 | 36 | 12
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group | Total
Number analyzed (Participants) | 36 | 36 | 12 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 8 | 52
  >=65 years | 13 | 15 | 4 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.7) | 63.3 (8.9) | 59.2 (9.1) | 62.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 9 | 41
  Male | 19 | 21 | 3 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 36 | 36 | 12 | 84

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sensory Nerve Block
Description: The primary outcome will be time to resolution of the nerve block as assessed by pinprick over the saphenous nerve distribution. Testing will occur every two hours.
Time Frame: 12 to 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
Number analyzed (Participants) | 36 | 36 | 12
hours | 37.00 (11.18) | 31.75 (10.50) | 29.67 (6.76)

2. Secondary Outcome: Verbal Pain Scores
Description: Verbal Pain Scores will be compared between groups as obtained every six hours during hospitalization. Patients will be asked to provide verbal pain scores both at rest and with movement on a scale of 0-10 (0 being no pain and 10 being the worst pain). These scores will be taken at 0, 6, 12, 18, 24, and 30 hours.
Time Frame: 0 to 30 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 4mg Perineural Dexamethasone: 4 mg of dexamethasone will be included in the saphenous nerve block mixture including 20 ml of 0.25% bupivacaine with 1:400,000 epinephrine. No systemic dexamethasone will be given.
  Resting pain score 0 hours post-op
- 1 mg Perineural Dexamethasone: 1 mg of dexamethasone will be included in the saphenous nerve block mixture including 20 ml of 0.25% bupivacaine with 1:400,000 epinephrine. No systemic dexamethasone will be given.
  Resting pain score 0 hours post-op
- Placebo: This group will receive only the saphenous nerve block mixture including 20 ml of 0.25% bupivacaine with 1:400,000 epinephrine. Dexamethasone will not be administered to this group systemically or perineural.
  Resting Pain score 0 hours post-op
Arm/Group | 4mg Perineural Dexamethasone | 1 mg Perineural Dexamethasone | Placebo
Number analyzed (Participants) | 36 | 36 | 12
units on a scale
  0h | 2.1 (2.5) | 2.3 (2.5) | 2.1 (2.4)
  6h | 0.8 (1.7) | 1.3 (2.3) | 1.1 (2.1)
  12h | 1.7 (1.8) | 2.1 (2.5) | 3.0 (2.6)
  18h | 1.6 (1.9) | 1.8 (2.1) | 3.3 (2.6)
  24h | 1.5 (1.7) | 1.8 (2.0) | 3.1 (2.0)
  30h | 2.4 (2.2) | 3.1 (2.7) | 4.3 (2.3)

3. Secondary Outcome: Rate of Post Operative Nausea and Vomiting
Description: Number of participants that experienced nausea and vomiting was recorded.
Time Frame: 0 to 30 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
Number analyzed (Participants) | 36 | 36 | 12
Participants | 5 | 14 | 4

4. Secondary Outcome: Neurologic Complications
Description: Each patient will be followed for neurologic complications (paresthesias, etc) if they should occur.
Time Frame: throughout study completion, up to 48 hours
Measure: Mean (Standard Deviation); unit: neurological complications
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
Number analyzed (Participants) | 36 | 36 | 12
neurological complications | 0 (0) | 0 (0) | 0 (0)

5. Secondary Outcome: Post Operative Opioid Use and Consumption
Description: Amount of opioid use and consumption was recorded.
Time Frame: 0-30 hours
Measure: Mean (Standard Deviation); unit: mg oxycodone equivalents
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
Number analyzed (Participants) | 36 | 36 | 12
mg oxycodone equivalents | 27.16 (24.35) | 26.04 (24.81) | 42.33 (26.30)

6. Secondary Outcome: Time to First Opioid Analgesic Request
Description: Time it took for the first opioid analgesic request was recorded.
Time Frame: 0 to 36 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
Number analyzed (Participants) | 36 | 36 | 12
minutes | 686.18 (420.41) | 654.97 (384.05) | 658.17 (424.66)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 72 hours post-operatively.
Arm/Group | 4 mg Perineural Dexamethasone Group | 1 mg Perineural Dexamethasone Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/12
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02462148/Prot_SAP_000.pdf